CLINICAL TRIAL: NCT01481636
Title: Association of Health Outcomes With Severity of OSA Symptomatology- a Correlation Study.
Brief Title: Assessing the Symptoms of Obstructive Sleep Apnea
Acronym: OSA
Status: Completed | Type: Observational
Sponsor: Bangor University (Other)
Responsible Party: Sponsor
Other Study IDs: REC No: 11/WNo:01/2; Earing 11/WNo01/2 (Other: North West Wales Research Ethics Committee)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; correlation; AHI; symptoms; mechanisms
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment, OSA (AHI >15): Patients with OSA recruited prior to receiving NHS treatment.

SUMMARY:
The purpose of this study is to investigate the correlation between health outcomes associated with the severity of obstructive sleep apnea (OSA) symptomatology, the findings will guide the design of interventional studies.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a condition characterised by periods of narrowing of the pharyngeal airways during sleep causing hypoxic and hypercapnic episodes with the cessation of ventilation. Considering the high number of overweight and obese individuals in Western society the understanding of the pathomechanisms behind OSA are important. This observational study aims to investigate the correlations between the severity of Obstructive Sleep Apnea assessed by the apnea-hypopnea index (AHI) and different health outcomes associated with the OSA.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≤39
* Not received any treatment for Obstructive Sleep Apnea.
* Is a non-smoker
* Is not epileptic
* Epworth Sleepiness Scale ≥ 10.
* Patient's on Statins or antihypertensive drugs are included as so frequent in OSA.

Exclusion Criteria:

* Body Mass Index ≥ 39.
* Presence of significant or unstable Renal, Liver or Heart Failure.
* Receiving anti-diabetic treatment.
* Is a smoker.
* Is epileptic
* Presence of significant or unstable psychological morbidities.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild to severe recently diagnosed Obstructive Sleep Apnea patients selected by physician who have not received any treatment for their condition. Selected from Ysbyty Gwynedd in North Wales.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | one night within four weeks of study.
  AHI refers to how is the number of apneas and hypopneas per an hour of sleep.

SECONDARY OUTCOMES:
Residual volume | Within four weeks of recruitment prior to CPAP treatment
  Volume of air remaining in lungs after full expiration
Functional residual volume | Within four weeks of recruitment prior to CPAP treatment
  Air present in lungs at the end of passive expiration
Total lung capacity | Within four weeks of recruitment prior to CPAP treatment
  Total volume of lungs
Forced Vital capacity | Within four weeks of recruitment prior to CPAP treatment
  Maximum amount of air which can be expired from the lungs following a full inspiration
Forced expiratory volume in one second (FEV1) | Within four weeks of recruitment prior to CPAP treatment
  Maximum amount of air which can be expired from the lungs in one second.
Airway Resistance | Within four weeks of recruitment prior to CPAP treatment
  Opposition of flow caused by forces of friction.
Plasma 2-arachidonoylglycerol (2-AG) | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment.
  Ligand of the G-protein coupled CB1 and CB2 receptors, has been found to be correlated with Oleylethanolamide (OEA) in OSA patients have various effects on energy metabolism.
Plasma Anandamide (ANA) | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  Ligand of the G-protein coupled CB1 and CB2 receptors, found to be correlated with blood pressure in OSA after the adjustment of confounding variables. Have various effects on energy metabolism.
Plasma oleoylethanolamine (OEA) | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  A lipid mediator which acts as an anorexigenic (appetite suppressant), and is elevated with sleep deprivation.
Plasma Leptin | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  Circulating protein produced in adipose tissue. Elevated in OSA and obesity. Leptin may reduce respiratory depression.
Plasma Adiponectin | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  Hormone secreted by adipocytes (Fat cells). Adiponectin is closely linked to metabolism and may have anti-inflammatory properties.
Plasma C-reactive Protein | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  Marker of inflammation.
Insulin | Within four weeks of recruitment prior to CPAP treatment and after four weeks of CPAP treatment
  Hormone which causes liver and muscle and fat cells to take up glucose to convert to glycogen. OSA is associated with insulin resistance.
Neck circumference | Within four weeks of recruitment prior to CPAP treatment
Waist circumference | Within four weeks of recruitment prior to CPAP treatment
Hip circumference | Within four weeks of recruitment prior to CPAP treatment
Weight | Within four weeks of recruitment prior to CPAP treatment
Fat-free mass | Within four weeks of recruitment prior to CPAP treatment
  Non-fat components of the human body estimated non-invasively using a bioimpedance measurement system.
Fat mass | Within four weeks of recruitment prior to CPAP treatment
  Fat components of the human body estimated non-invasively using bioimpedance measurement system.
Maximal Inspiratory pressure | Within four weeks of recruitment prior to CPAP treatment
  Measured at residual volume, reflects the strength of the diaphragm and other inspiratory muscles.
Rate of inspiratory muscle fatigue | Within four weeks of recruitment prior to CPAP treatment
  The decline in maximal inspiratory pressure following inspiration against a resistance.
Chest RPE | Within four weeks of recruitment prior to CPAP treatment
  Rating of perceived exertion in the chest and associated airways during the inspiratory fatigue protocol.
Dyspnea | Within four weeks of recruitment prior to CPAP treatment
  Rating of breathlessness half way through fatigue protocol and at the end of protocol.
Ventilation with 25% O2/ 6% CO2 | Within four weeks of recruitment prior to CPAP treatment
  Measures the breathing response to high oxygen and high CO2 therefore assessing the central chemoreceptors response only.
Ventilation with 13% O2 | Within four weeks of recruitment prior to CPAP treatment
  Measures the breathing response to low oxygen. Designed to Assess the response to the peripheral chemoreceptors.
Ventilation with 13% O2 / 6% CO2 | Within four weeks of recruitment prior to CPAP treatment
  Measures the breathing response to low oxygen and high CO2. Designed to assess the response of the sum of the peripheral and central chemoreceptors
Mean RR interval | Within four weeks of recruitment prior to CPAP treatment
  Time domain measure: Average time interval between the heart beats R waves
SDNN | Within four weeks of recruitment prior to CPAP treatment
  Time domain measure: The standard deviation of all RR intervals
NN50 count | Within four weeks of recruitment prior to CPAP treatment
  Time domain measure: The number of pairs of adjacent RR intervals differing by more than 50 ms in the entire analysis interval.
NN50 of total HR (%) | Within four weeks of recruitment prior to CPAP treatment
  Time domain measure: NN50 count divided by total number of all RR intervals.
HRV triangular index | Within four weeks of recruitment prior to CPAP treatment
  The total number of RR intervals divided by maximum height of the histogram excluding boundaries.
Low frequency domain | Within four weeks of recruitment prior to CPAP treatment.
  Frequency domain analysis: represents 0.04-0.15 Hz reflecting sympathetic activity.
High frequency domain | Within four weeks of recruitment prior to CPAP treatment.
  Frequency domain analysis: represents 0.15-0.40 Hz reflecting parasympathetic activity.
LF/HF ratio | Within four weeks of recruitment prior to CPAP treatment.
  The ratio of low frequency (0.04 - 0.15 Hz) to high (0.15-0.40 Hz) frequency recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher MN Earing, MSc, Principal Investigator — School of Sport, Health and Exercise Sciences, Bangor University
Locations (1):
- Betsi Cadwaladr University Health Board, Bangor, Gwynedd, United Kingdom